CLINICAL TRIAL: NCT07368036
Title: MR 7700 Multinuclear Application Clinical Study
Brief Title: MR 7700 Multinuclear Application Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 300957
Record Dates: First submitted 2025-12-01; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: MR Multinuclear; Image Quality; Device Convenience; Device Stability; System Safety
Keywords: multinuclear; MR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Experimental)
  Interventions: Device: MR Scanning with Phosphorus nucleus + Sodium nucleus
- Patient (Experimental)
  Interventions: Device: MR Scanning with Phosphorus nucleus + Sodium nucleus

INTERVENTIONS:
Device: MR Scanning with Phosphorus nucleus + Sodium nucleus — Using the Magnetic Resonance Equipment to perform phosphorus nucleus (31P) and sodium nucleus (23Na) scanning

SUMMARY:
The purpose of this clinical trial is to use the medical magnetic resonance imaging system MR 7700 to perform phosphorus (31P) and sodium (23Na) scanning imaging on the human body, evaluate the image quality of phosphorus (31P) and sodium (23Na) scanning, as well as the machine convenience, machine stability, and system safety of the entire system.

ELIGIBILITY:
Inclusion Criteria:

* • 18 ≤ Age ≤ 75 years old;

  * Clear mind, able to cooperate, and capable of autonomous behavior;
  * Voluntarily agree to participate in this clinical trial and sign the informed consent form for the subjects

Exclusion Criteria:

* • Individuals with claustrophobia.

  * On the day of scanning, the subject's body temperature was above 39.5 ℃.
  * Plan to become pregnant, pregnant, and breastfeeding women within 6 months.
  * Other implants, prostheses, foreign bodies, patches, etc. that are not suitable for magnetic resonance imaging examination; There are electronic implants such as pacemakers, stimulators, insulin pumps, cochlear implants, etc.
  * Critical patients equipped with various rescue devices, as well as subjects with any emergency medical conditions requiring first aid.
  * Subjects with poor compliance, which the researchers believe should be excluded.
  * Other situations that the investigators believe are not suitable for participating in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The excellent and good rate of Spectral image quality of 31P-MRS | 14 days (anticipated) after finishing 31P-MRS scanning
  Spectral image quality of phosphorus nucleus (31P) in each site (muscle, liver, heart)，will be assessed by Likert score (1-5) .
  The final evaluation of image quality at 3 points or above is considered excellent and good.The rate of excellent and good should be over 75%.
The excellent and good rate of image quality of 23Na-MRI | 14 days (anticipated) after finishing 23Na-MRI scanning
  Image quality of sodium nuclei (23Na) in each site (liver, cartilage), will be assessed by Likert score (1-5) . The final evaluation of image quality at 3 points or above is considered excellent and good.The rate of excellent and good should be over 75%.

SECONDARY OUTCOMES:
The Device convenience of the entire system | 14 days (anticipated) after finishing scanning
  A three-scale assessment will be used for evaluate the device convenience of the entire system from the aspects of subject positioning, scanning interface, scanning sequence, image processing, microphone communication, and image storage/transmission and management.
  A three-scale criteria- Satisfied, General, Dissatisfied Assessment criteria: The parameters should all reach "General or Satisfied", indicating that the case meet the device convenience.
Device stability | 14 days (anticipated) after finishing scanning
  Evaluate the stability of the device from the aspects of system startup, system shutdown, abnormal interruption during scanning, image display after scanning, and missing image reconstruction.
  A three-scale criteria- Satisfied, General, Dissatisfied. Assessment criteria: The parameters should all reach "General or Satisfied", indicating that the case meet the device stability.
System security | 14 days (anticipated) after finishing scanning
  The technician observes whether there are any system safety issues during the scanning of each image instance After the scan, a "yes" or "no" judgment is made based on the occurrence of each assessment item. If all assessment items are rated as "none", it indicates that the system is safe.
Adverse event | From the time the subjects signed the ICF to completion of study visit(1 day).
  Analyze the adverse events during the clinical trial process, summarize and analyze the frequency and percentage of all adverse events (including serious adverse events) in a list, and classify them based on their correlation with the device.

IPD SHARING:
Plan to Share IPD: Undecided